CLINICAL TRIAL: NCT06119152
Title: Digital Equity for Stroke Approach Pilot Study
Brief Title: Digital Equity for Stroke Approach
Acronym: DESA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1849255-4
Record Dates: First submitted 2023-07-11; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Blood Pressure, High
Keywords: Telehealth; Digital Health; Remote Device Monitoring; Health Disparities; Afro-Caribbean
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- Intervention (Experimental): The DESA Intervention will use a telehealth device to help the patient take blood pressure daily, and monitor blood pressure management.
  Interventions: Behavioral: DESA

INTERVENTIONS:
Behavioral: DESA — Intervention group is monitored via remote bp monitoring and telehealth device.
  Arms: Intervention

SUMMARY:
A community-academic partnership composed of a State University of New York (SUNY) Downstate Health Sciences University inter-disciplinary team of scientists (representing public health, medical informatics, vascular neurology/stroke center) and the Digital Equity Community Advisory Board (DECA) will guide our research. This is an NIH R21 pilot study. Our Specific Aims are designed to inform the sample design and research priorities for a larger NIH R01 experimental study and to serve as a platform for similar studies with other health conditions. We propose a mixed-methods study design with the following aims:

1. Assess and build setting, community, and user fit of DESA, leveraging qualitative methods and simulation telehealth encounters between the patient and neurologist.
2. Conduct a 9-month pilot randomized control trial (RCT) of DESA in a Central Brooklyn stroke population to examine the feasibility and preliminary efficacy. We will randomize 50 adults to DESA and 30 to usual care. The primary outcome will be BP control. Secondary outcomes include the number of BP measurements and medication compliance. Our primary hypothesis is that patients randomized to the DESA will significantly reduce systolic blood pressure at 9 months.
3. Examine barriers and facilitators to the adoption and integration of DESA into routine stroke care utilizing key informant interviews and user satisfaction surveys with neurologists and intervention participants.

ELIGIBILITY:
Inclusion Criteria:

* African American or Afro-Caribbean
* 18 years or over
* Experienced a stroke in the last 6 years
* A score between 2 and 4 on the Modified Rankin Scale2
* Has a formal or informal caregiver (e.g., relative, health aide or other) to assist them in activities of daily living
* Has a primary care physician at University Hospital of Brooklyn (UHB)

Exclusion Criteria:

* Mental illness (severe depression)
* dementia
* Non-English speakers
* aphasia
* severe dysarthria (slurred speech/impediment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Change | 9 months
  Blood Pressure (Systolic and Diastolic) will be recorded by telehealth device daily

SECONDARY OUTCOMES:
Number of Blood Pressure readings/week | 9 months
  Blood Pressure (Systolic and Diastolic) will be recorded by telehealth device daily, so days measured are received from this.
Medication Adherence | 9 months
  Measured by medication adherence survey, at beginning, midpoint, and endpoint of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: David R Kaufman, PhD, FACMI, Principal Investigator — SUNY Downstate Health Sciences University; Aimee Afable, PhD, MPH, Principal Investigator — SUNY Downstate Health Sciences University
Locations (1):
- University Hospital at Downstate, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No